CLINICAL TRIAL: NCT02561923
Title: Randomized, Parallel-Group, 2-Part Study to Assess the Independent Effects of 4-Factor Prothrombin Complex Concentrate and Tranexamic Acid on Bleeding Parameters and Pharmacodynamics After a Punch Biopsy Procedure in Healthy Subjects Treated With Rivaroxaban
Brief Title: A Study to Assess the Independent Effects of 4-Factor Prothrombin Complex Concentrate and Tranexamic Acid on Bleeding/Pharmacodynamics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107832; 39039039NAP1004 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2015-08-21; First posted 2015-09-28 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Rivaroxaban; XARELTO
MeSH Terms: interventions — Rivaroxaban; Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rivaroxaban (Experimental): Participants will be administered a single 20 milligram (mg) dose of rivaroxaban orally on Day 1 in Part 1.
  Interventions: Drug: Rivaroxaban
- Rivaroxaban plus tranexamic acid (TXA) (Experimental): Participants will be administered rivaroxaban (20 mg every 12 hrs) on Days 1 through 3 and a single 20 mg dose will be given on the morning of Day 4, all doses given orally. Following rivaroxaban adminsitration on Day 4, tranexamic acid (TXA) 1.0 gram (g) - (over 10 mins) intravenously administered on Day 4 in Part 2.
  Interventions: Drug: Rivaroxaban; Drug: Tranexamic acid
- Rivaroxaban plus Kcentra (Experimental): Participants will be administered rivaroxaban (20 mg every 12 hrs) on Days 1 through 3 and a single 20 mg dose will be given on the morning of Day 4, all doses given orally. Following rivaroxaban adminsitration on Day 4, participants will be randomized to receive a single dose of Kcentra (a 4-factor PCC), 50 international units per kilogram (IU/kg), intravenously administered (maximum rate of 210 [international units per minute] IU/min) on Day 4 in Part 2.
  Interventions: Drug: Rivaroxaban; Drug: Kcentra, a 4-factor PCC
- Rivaroxaban plus Saline (Experimental): Participants will be administered rivaroxaban (20 mg every 12 hrs) on Days 1 through 3 and a single 20 mg dose will be given on the morning of Day 4, all doses given orally. Following rivaroxaban adminsitration on Day 4, saline [Kcentra saline control or TXA saline control] on Day 4 in Part 2.
  Interventions: Drug: Rivaroxaban; Drug: Saline

INTERVENTIONS:
Drug: Rivaroxaban — A single dose of 20 milligram (mg) of rivaroxaban orally will be administered to participants on Day 1 in part 1 and through day 1 and 3 with a final 20 mg dose administered on the morning of Day 4 in part 2.
Drug: Tranexamic acid — 1.0 g single dose of tranexamic acid (TXA), intravenously administered (over 10 mins) on Day 4.
  Arms: Rivaroxaban plus tranexamic acid (TXA)
Drug: Kcentra, a 4-factor PCC — Kcentra, a 4-factor PCC, 50 IU/kg, single dose, intravenously administered (maximum rate of 210 [international units] IU/min) on Day 4.
  Arms: Rivaroxaban plus Kcentra
Drug: Saline — Saline [Kcentra saline control or TXA saline control] on Day 4.
  Arms: Rivaroxaban plus Saline

SUMMARY:
The purpose of this study is to assess the independent effects of both a 4-Factor prothrombin complex concentrate (PCC) - (Kcentra) and Tranexamic acid (TXA) on the bleeding parameters (bleeding duration and blood volume) following a punch biopsy, in addition to assessing their effects on the anticoagulant/pharmacodynamic (prothrombin time and endogenous thrombin potential) changes induced by rivaroxaban at steady state, to better understand their potential role in bleeding reversal.

DETAILED DESCRIPTION:
This is a 2 part, single center study to be conducted in healthy men and women. Part 1 (open-label) consists of Screening Phase (within 28 days before admission into the study center on Day -1), followed by a 3 day treatment period and a follow-up visit on Day 8. A single oral 20 milligram (mg) dose of rivaroxaban will be administered on Day 1. Pharmacokinetic (PK), pharmacodynamics (PD), and punch biopsy parameters will be assessed. Part 2 (double-blind) consists of Screening Phase (within 28 days before admission into the study center on Day -1), followed by a 8 day treatment period (Day -1 to Day 7) and a follow-up visit on Day 11. Rivaroxaban (20 mg every 12 hrs) will be administered on Days 1 through 3 and single 20 mg dose will be given on the morning of Day 4. A single dose of either 4-factor PCC, TXA or saline (Placebo) will be administered in a randomized, blinded fashion on Day 4. PK, PD, Exploratory Bio-markers and punch biopsy parameters will be assessed. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight kilogram [kg]/height^2 meters [m]^2) between 18 and 30 kg/m2 (inclusive), and body weight between 50 and 100 kg;
* Participants must have coagulation test results of prothrombin time (PT) and a partial thromboplastin time (PTT) within normal limits at Screening
* Must have normal renal function, as per medical history
* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (eg, double-barrier method or male partner sterilization) before entry and throughout the study. (Note: combined hormonal contraception should not be used)
* Non-smoker (Note: subjects should not have used nicotine-containing products within 30 days before study drug administration)
* If a woman, must have a negative serum Beta-human chorionic gonadotropin (hCG)] pregnancy test at Screening; and a negative serum pregnancy test on Day -1 of the study
* If a man, must agree to use adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease (including history of definite myocardial infarction, cerebrovascular accident, percutaneous transluminal coronary angioplasty or coronary artery bypass graft within 6 months before the Screening visit, or a previous intracranial hemorrhage at any time, known history of lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, seizure disorder, infection, skin disease, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results
* Participants with any history of thrombosis, inherited or acquired thrombophilia, bleeding diathesis or coagulopathy (including any abnormal bleeding or blood dyscrasias), hematologic disease, clinically significant hemorrhagic disorder, excessive bruising, bleeding from nose or gums or known disorders with increased bleeding risk (eg, acute gastritis, acute peptic ulcer), serious bleeding including gastrointestinal bleeding requiring hospitalization, intracranial bleeding of any type, or uncontrollable postoperative bleeding
* Known antithrombin III, Protein C, or Protein S deficiency, Factor V Leiden or prothrombin gene 20210 mutation, anticardiolipin (immunoglobulin G [IgG] and immunoglobulin M [IgM]) or antiphospholipid antibodies, or family history of unexplained thrombotic disorders
* History of intracranial tumor or aneurysm or known abdominal aneurysm
* Clinically significant abnormal physical examination, vital signs or 12-lead electrocardigram [ECG] at Screening or at admission to the study center on Day -1, as deemed appropriate by the investigator. This would include: resting pulse >100 or <40 beats per min, blood pressure systolic >140 or <90 millimeters per mercuric level [mmHg], and diastolic blood pressure > 90 or < 50 mmHg (pulse and blood pressure measurements should be taken in a supine position, after resting for at least 5 minutes)
* Participants for whom surface blood vessels could not be visualized, or who have a history of likelihood of forming keloid scars
* Use of any prescription or nonprescription medication (including antiplatelet, anticoagulants, aspirin, non-steroidal anti-inflammatory drugs, vitamins and herbal supplements), within 7 days before the first dose of the study drug is scheduled
* Known allergy to the study drugs or any of the excipients of the formulations
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-06-17 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Blood Volume in Part 1 | Day-1 (Baseline) and 4 hour (hr) postdose on Day 1
  Volume of blood (BV) collected after a punch biopsy is performed.
Change From Baseline in Bleeding Duration in Part 1 | Day-1 (Baseline) and 4 hr postdose on Day 1
  Bleeding duration (BD) after a punch biopsy is performed.
Mean Change in Thrombin Generation Assay (TGA) - Endogenous Thrombin Potential (ETP) Lag-time in Part 2 | Predose (Baseline) and up to 72 hrs postdose on Day 4
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in lag time (time required until thrombin is generated) will be observed.
Mean Change in Thrombin Generation Assay (TGA) - Endogenous Thrombin Potential (ETP) Peak in Part 2 | Predose (Baseline) and 72 hours postdose on Day 4
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in peak (the maximal effect on thrombin generation) will be observed.
Mean Change in Thrombin Generation Assay (TGA) - Endogenous Thrombin Potential (ETP) Time to Peak in Part 2 | Predose (Baseline) and 72 hours postdose on Day 4
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in time-to-peak (time required to reach maximal effect on thrombin generation) will be observed.
Mean Change in Thrombin Generation Assay (TGA) - Endogenous Thrombin Potential (ETP) Area Under Curve (AUC) in Part 2 | Predose (Baseline) up to 72 hours on Day 4
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in AUC (the overall effect on thrombin generation) will be observed.
Mean Change in Prothrombin Time (PT) in Part 2 | Predose (Baseline) up to 72 hours on Day 4
  Prothrombin Time is a global clotting test that is used for the assessment of the extrinsic pathway of the blood coagulation cascade.
Change From Baseline in Blood Volume in Part 2 | Predose (Baseline) and 72 hours on Day 4
Change From Baseline in Bleeding Duration in Part 2 | Predose (Baseline) and 72 hours on Day 4

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) in Part 1 | Predose and up to 24 hrs postdose on Day 1
Time to Maximum Observed Plasma Concentration in Part 1 (Tmax) | Predose and up to 24 hrs post-dose
Area under Plasma Concentration Time Curve From Time 0 to 24 in Part 1 (AUC [0 TO 24] | Predose and up to 24 hrs postdose on Day 1
Maximum Observed Plasma Concentration (Cmax) in Part 2 | Predose and up to 72 hrs postdose on Day 4
Minimum Observed Plasma Concentration (Cmin) in Part 2 | Predose Days 1 to 4
Time to Maximum Observed Plasma Concentration (Tmax) in Part 2 | Predose and up to 72 hrs postdose on Day 4
Area under plasma concentration time curve during the dosing interval (AUCtau) in Part 2 | Predose and up to 24 hours
Mean Change in Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP) Lag-time in Part 1 | Predose (Baseline) up to 24 hours on Day 1
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in lag time (time required until thrombin is generated) will be observed.
Mean Change in Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP) Peak in Part 1 | Predose (Baseline) up to 24 hours on Day 1
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in peak (the maximal effect on thrombin generation) will be observed.
Mean Change in Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP) Time to Peak in Part 1 | Predose (Baseline) up to 24 hours on Day 1
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in time-to-peak (time required to reach maximal effect on thrombin generation) will be observed.
Mean Change in Thrombin Generation Assay (TGA) Endogenous Thrombin Potential (ETP) Area Under Curve (AUC) in Part 1 | Predose (Baseline) up to 24 hours on Day 1
  The thrombin generation assay (TGA) is based on the premise that measurements of thrombin generation are indicative of the overall coagulating capacity of the individual. The data derived from the thrombography can be used to determine the ETP, which in turn provides a functional assessment of the overall clotting cascade. Change in AUC (the overall effect on thrombin generation) will be observed.
Mean Change in Prothrombin Time (PT) in Part 1 | Predose (Baseline) up to 24 hours on Day 1
  Prothrombin Time is a global clotting test that is used for the assessment of the extrinsic pathway of the blood coagulation cascade.
Trough Plasma Concentration (Ctrough) in Part 2 | Predose and up to 72 hrs postdose on Day 4
  Ctrough is the trough plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 37 Days (Part 1) and Up to 40 Days (Part 2)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- Overland Park, Kansas, United States

REFERENCES:
- See also: Randomized,Parallel-Group,2-Part Study to Assess the Independent Effects of 4-Factor Prothrombin Complex Concentrate and Tranexamic Acid on Bleeding Parameters and Pharmacodynamics After Punch Biopsy Procedure in Healthy Subjects Treated With Rivaroxaban — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=10698&filename=CR107832_CSR.pdf